CLINICAL TRIAL: NCT00790530
Title: Automated Telephone Outreach With Speech Recognition to Improve Diabetes Care: A Randomized Controlled Study
Acronym: ATO-SR-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Steven R. Simon, Principal Investigator, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1-05-JF-40
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Information Technology; Health Plans
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATO-SR (Experimental): Automated Telephone Outreach with Speech Recognition
  Interventions: Behavioral: Automated Telephone Outreach with Speech Recognition
- Usual Care (No Intervention): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Automated Telephone Outreach with Speech Recognition — Automated Telephone Outreach with Speech Recognition
  Arms: ATO-SR
Other: Usual Care — Usual Care
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate the effectiveness of automated telephone outreach with speech recognition to improve diabetes care.

DETAILED DESCRIPTION:
Randomly allocate a total of 1200 health plan members with diabetes to automated telephone outreach with speech recognition (ATO-SR; N = 600) or usual care (N = 600). The intervention is a series of three calls, using automated calls, originating from the health plan, using interactive speech recognition technology, spaced approximately 4-6 weeks apart, to encourage participants to fulfill the recommended testing (dilated eye examinations, glycated hemoglobin, LDL-cholesterol, microalbumin) that had not been performed received in the preceding year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diabetes, defined as either 1) filled a prescription for insulin or an oral hypoglycemic agent; or, 2) had two outpatient or one inpatient or two outpatients encounter claims with an ICD9-CM or CPT code indicating diabetes.
* Gap in a key diabetes management metric as evidenced by no claim for a dilated eye examination in the prior 15 months and no claim for one or more of the following tests: glycated hemoglobin, LDL-cholesterol, or microalbumin. (Individuals with evidence of having received ACE-inhibitors or angiotensin receptor blockers were considered to have had a microalbumin test.)

Exclusion Criteria:

* No primary care clinician in the data base
* Those who had previously asked the health plan to exclude them from research or quality improvement
* Women whose claim records contained diagnoses suggesting gestational diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2006-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Completion of dilated eye examination | 12-months following intervention

SECONDARY OUTCOMES:
Completion of glycated hemoglobin testing (HbA1c) | one-year following intervention
Completion of LDL-cholesterol testing | one year following intervention
Completion of microalbumin testing | one-year following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Simon, MD, Principal Investigator — Harvard Pilgrim Health Care
Locations (1):
- Harvard Pilgrim Health Care, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Simon SR, Trinacty CM, Soumerai SB, Piette JD, Meigs JB, Shi P, Ensroth A, Ross-Degnan D. Improving diabetes care among patients overdue for recommended testing: a randomized controlled trial of automated telephone outreach. Diabetes Care. 2010 Jul;33(7):1452-3. doi: 10.2337/dc09-2332. Epub 2010 Mar 31. PMID 20357376